CLINICAL TRIAL: NCT04780724
Title: Evaluation of SpO2 Measurement Using a Smartwatch
Acronym: ESMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: smartwatch21
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Hypoxia; Hypercapnia
Keywords: SpO2; pulse oximetry; smartwatch
MeSH Terms: conditions — Hypoxia; Hypercapnia | interventions — nitrox

STUDY DESIGN:
Intervention Model Description: All participants go through all study arms, in random order. Two measuring devices are active simultaneously during measurement on each participant and their functioning is compared.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoxic (Experimental): Participants inhale ambient air, the hypoxic gas mixture, and ambient air.
  Interventions: Other: Hypoxic gas mixture; Other: SpO2 measurement
- Hypercapnic (Experimental): Participants inhale ambient air, the hypercapnic and hypoxic gas mixture, and the ambient air.
  Interventions: Other: Hypercapnic and hypoxic gas mixture; Other: SpO2 measurement

INTERVENTIONS:
Other: Hypoxic gas mixture — Gas mixture of 12% O2 and 88% N2 for five minutes.
  Arms: Hypoxic
Other: Hypercapnic and hypoxic gas mixture — Gas mixture of 12% O2, 5% CO2, and 88% N2 for five minutes.
  Arms: Hypercapnic
Other: SpO2 measurement — Two SpO2 measuring devices are active simultaneously during measurement.

SUMMARY:
The aim of the study is to compare the measurement of peripheral blood oxygen saturation using a smartwatch with a medical-grade pulse oximeter.

DETAILED DESCRIPTION:
Recently, wearables, like smartwatches, have been gaining new possibilities in monitoring biological signals and they are used for home monitoring of health conditions. The newest models of smartwatches even measure peripheral blood oxygen saturation (SpO2). The study aims to compare the measurement of peripheral blood oxygen saturation using the latest smartwatch with a medical-grade pulse oximeter under the condition of normobaric hypoxia. Healthy participants will breathe oxygen-reduced mixtures (the hypoxic gas mixture of 12% O2 and 88% N2 and the hypercapnic and hypoxic gas mixture of 12% O2, 5% CO2, and 83% N2), which will temporarily reduce their blood oxygen saturation. SpO2 measurements will be taken by hand from the watch and the pulse oximeter simultaneously. The agreement of the measurements of both devices will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers from the Czech Technical University

Exclusion Criteria:

* pregnancy
* severe cardiovascular conditions
* severe asthma or other severe respiratory conditions
* injury to the upper limbs or hands that could affect the peripheral perfusion
* diabetes
* hypotension or hypertension

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Similarity of SpO2 readings | 2 hours
  The agreement of SpO2 measurements of both monitoring devices will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Rafl Huttova, Principal Investigator — Czech Technical University in Prague
Locations (1):
- Faculty of Biomedical Engineering, Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafl J, Kulhanek F, Kudrna P, Ort V, Roubik K. Response time of indirectly accessed gas exchange depends on measurement method. Biomed Tech (Berl). 2018 Nov 27;63(6):647-655. doi: 10.1515/bmt-2017-0070. PMID 28802098
- [Background] Lauterbach CJ, Romano PA, Greisler LA, Brindle RA, Ford KR, Kuennen MR. Accuracy and Reliability of Commercial Wrist-Worn Pulse Oximeter During Normobaric Hypoxia Exposure Under Resting Conditions. Res Q Exerc Sport. 2021 Sep;92(3):549-558. doi: 10.1080/02701367.2020.1759768. Epub 2020 Jul 7. PMID 32633688
- [Derived] Rafl J, Bachman TE, Rafl-Huttova V, Walzel S, Rozanek M. Commercial smartwatch with pulse oximeter detects short-time hypoxemia as well as standard medical-grade device: Validation study. Digit Health. 2022 Oct 11;8:20552076221132127. doi: 10.1177/20552076221132127. eCollection 2022 Jan-Dec. PMID 36249475